CLINICAL TRIAL: NCT01714284
Title: Multicenter Randomized Clinical Study Evaluating the Efficacy of Dietary Intervention and Weight Loss in Improving Psoriasis
Brief Title: Efficacy Study of Dietary Intervention and Weight Loss in Improving Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Studi Gised (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSODIET1
Record Dates: First submitted 2012-10-23; First posted 2012-10-25 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Psoriasis
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet and Exercise (Experimental)
  Interventions: Behavioral: Diet and Exercise
- Informative (Sham Comparator)
  Interventions: Behavioral: Informative

INTERVENTIONS:
Behavioral: Informative — The intervention consists in a simple informative counseling about the utility of weight loss for clinical control of psoriatic disease.
  Other Names: informative, weight loss
  Arms: Informative
Behavioral: Diet and Exercise — The intervention consists in a 20 weeks quantitative and qualitative dietary plan for weight loss associated with physical exercise. The plan will be developed with the help of qualified staff (Dieticians) and elaborated in relation to individual needs of the patient.
  Other Names: diet, weight loss, exercise
  Arms: Diet and Exercise

SUMMARY:
This is a multicenter randomized controlled clinical trial evaluating the impact of a structured non pharmacological intervention consisting in intensive weight reduction (qualitative and quantitative changes in diet associated with physical exercise) compared to an intervention based on a simple informative counseling about the utility of weight loss for clinical control of psoriatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic plaque psoriasis
* BMI > 25 Kg/m²
* Patients under systemic treatments for psoriasis or candidates for such treatments

Exclusion Criteria:

* Diagnosis of other type of psoriasis or psoriatic arthritis
* Patients under local treatments or candidates for such treatments
* Patients expected to have poor compliance at follow-up evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Any change from baseline of PASI index | 20 weeks

SECONDARY OUTCOMES:
Percent change from baseline of PASI index equal to or greater than 50% (PASI50+) | 8 weeks, 16 weeks, 20 weeks
Percent change from baseline of PASI index equal to 100% (PASI100) | 8 weeks, 16 weeks, 20 weeks
Any change from baseline of PASI index | 8 weeks, 16 weeks, 20 weeks
Any reduction from baseline of Body Mass Index (BMI) | 8 weeks, 16 weeks, 20 weeks
Any reduction from baseline of waist circumference | 8 weeks, 16 weeks, 20 weeks
Percent change from baseline of PASI index equal to or greater than 75% (PASI75+) | 8 weeks, 16 weeks, 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Naldi, MD, Study Director — Centro Studi Gised; Alberto Giannetti, MD, Principal Investigator — University General Hospital of Modena
Locations (11):
- Italy (11):
  - Department of Dermatology; Bellaria-Maggiore Hospital, Bologna, Emilia-Romagna
  - Department of Dermatology; S.Orsola-Malpighi General Hospital, Bologna, Emilia-Romagna
  - Dermatology Department; M. Bufalini Hospital, Cesena, Emilia-Romagna
  - Department of Dermatology; S. Anna University Hospital, Ferrara, Emilia-Romagna
  - Department of Dermatology; G.B.Morgagni-L.Pierantoni Hospital, Forlì, Emilia-Romagna
  - Department of Dermatology; University General Hospital of Modena, Modena, Emilia-Romagna
  - Department of Dermatology; University General Hospital of Parma, Parma, Emilia-Romagna
  - Department of Dermatology; Hospital of Piacenza, Piacenza, Emilia-Romagna
  - Department of Dermatology; AUSL of Ravenna, Ravenna, Emilia-Romagna
  - Department of Dermatology; S. Maria Nuova Hospital, Reggio Emilia, Emilia-Romagna
  - Department of Dermatology; Infermi Hospital, Rimini, Emilia-Romagna